CLINICAL TRIAL: NCT00211367
Title: Treatment of Radiation Retinopathy With Open-Label Anecortave Acetate Sterile Suspension (15 mg)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: poor enrollment
Sponsor: Manhattan Eye, Ear & Throat Hospital (Other)
Collaborators: Alcon Research (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AA in Rad.Ret.
Expanded Access: Available
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2007-06-21 (Estimated); Status verified 2007-06

CONDITIONS: Eye Injuries
Keywords: Radiation Retinopathy
MeSH Terms: conditions — Eye Injuries | interventions — anecortave acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Anecortave Acetate

SUMMARY:
Radiation retinopathy is a disease of the retina. It occurs in people who have received or been exposed to radiation near the eyes. The blood vessels are abnormal and may grow which lead to scarring and a loss of central vision. Currently, the treatment for radiation retinopathy is laser photocoagulation. This treatment has been found to have limited use in this type of condition. Compassionate use of anecortave acetate injection is being considered to prevent the growth of the blood vessels under the retina.

DETAILED DESCRIPTION:
Patients will receive an injection of 15 mg of Anecortave acetate behind the eye to be treated ("study eye"). They will be evaluated every six months to determine if their condition is stable or worse. Following the injection of study medication, patients will not be required to come in to see the study physician. The investigator or study staff will call the patients on the day following injection to make sure there were no adverse effects to the injection. Patients will then come in for a Month 1 and a Month 3 follow-up visit. At the Month 3 follow-up visit, if patients are not showing stability or improvement, they may be offered either thermal laser or Photodynamic Therapy. They will remain in the study and remain eligible for a repeat injection of Anecortave Acetate at the Month 6 visit.

Patients will then been seen at Month 6 for a Re-treatment Evaluation Visit. If their condition is stable, they will be offered re-injection with the same study medication they received earlier. If Patients are not showing stability or improvement at the Month 6 visit, they may be offered thermal laser or Photodynamic Therapy in conjunction with the Anecortave Acetate injection.

Patients will then come back again for a Month 1 and a Month 3 visit and an Exit Visit, if necessary. If the patient's condition is worse, patients will be exited from this study and offered standard treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of radiation retinopathy.
2. Patients must be 18 years of age or older to receive treatment.
3. Visual acuity of 20/30 to 20/320 in study eye on the Early Treatment of Diabetic Retinopathy Study (ETDRS) visual acuity chart
4. Visual acuity of 20/800 or better in fellow eye on the ETDRS visual acuity chart.

Exclusion Criteria:

1. Patient with significantly compromised visual acuity in the study eye due to concomitant ocular conditions.
2. Patients who have undergone intraocular surgery within the last 2 months
3. Patient participating in any other investigational drug study.
4. Use of an investigational drug or treatment related or unrelated to their condition within 30 days prior to receipt of study medication.
5. Inability to obtain photographs to document choroidal neovascularization (CNV) (including difficulty with venous access)
6. Patient with significant liver disease or uremia.
7. Patient with known adverse reaction to fluorescein and indocyanine green or iodine.
8. Patient has a history of any medical condition which would preclude scheduled visits or completion of study
9. Patient has had insertion of scleral buckle in the study eye
10. Patient has received radiation treatment
11. Patient is on anticoagulant therapy with the exception of aspirin
12. Patient is pregnant or nursing.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2004-04; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
to investigate the use of anecortave acetate in radiation retinopathy | 24 months

SECONDARY OUTCOMES:
mean change of ETDRS VA from baseline to 24 monthe | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence A. Yannuzzi, MD, Principal Investigator — Manhattan Eye, Ear & Throat Hospital
Locations (1):
- Manhattan Eye, Ear & Throat Hospital, New York, New York, United States